CLINICAL TRIAL: NCT06415656
Title: Digital Multi-Vital Sign Monitoring for Early Detection of Cytokine Release Syndrome From Bispecific T-Cell Engagers and Chimeric Antigen Receptor Therapy
Brief Title: VitalTraq for the Detection of CRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Blue Spark Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00115012
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with hematologic malignancies (Experimental): Patients who are scheduled to receive CAR-T or BiTE through the Duke Adult Blood and Bone Marrow Transplant (ABMT) and Hematologic Malignancies Program.
  Interventions: Device: TempTraq; Device: VitalTraq

INTERVENTIONS:
Device: TempTraq — TempTraq (Blue Spark Technologies, Westlake, OH) is an FDA 510K cleared wearable, wireless temperature monitoring patch designed to continuously monitor and track body temperature.
Device: VitalTraq — VitalTraq (Blue Spark Technologies, Westlake, OH) is an experimental and novel multi-vital sign monitoring platform that allows for interval measurements of heart rate, heart rate variability, and blood pressure.

SUMMARY:
The purpose of this study is to evaluate two vital sign monitoring devices, TempTraq and VitalTraq, in patients with hematologic malignancies undergoing therapy with Chimeric antigen receptor T-cell therapy (CAR-T) or Bispecific T-cell engagers (BiTE) products. TempTraq is an axillary patch that is worn on the skin and continuously monitors a patient's body temperature. VitalTraq is a smartphone application that utilizes remote photoplethysmography technology via a 30-second facial scan to estimate the patient's blood pressure (BP), heart rate (HR), heart rate variability (HRV), and respiratory rate. These remote vital sign monitoring devices have the potential to promote earlier detection and intervention of treatment-related toxicities, including cytokine release syndrome (CRS) and febrile neutropenia.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at or over the age of 18 with hematologic malignancies undergoing treatment with chimeric antigen receptor (CAR) T-cell therapy or bispecific T-cell engagers (BiTE), as follows:

   * Axicabtagene ciloleucel
   * Lisocabtagene maraleucel
   * Brexucabtagene autoleucel
   * Idecabtagene vicleucel
   * Ciltacabtagene autoleucel
   * Obecabtagene autoleucel
   * Tisagenlecleucel
   * Blinatumomab
   * Mosunetuzumab
   * Talquetamab
   * Elranatamab
   * Teclistamab
   * Glofitamab
2. Owns a smart phone (e.g., iPhone, Android, Samsung) that is compatible with the VitalTraq app and that can connect to wi-fi. This will be assessed at screening.
3. Able to read and understand English
4. Willing and able to provide informed consent to the study

Exclusion Criteria:

1. Receiving a non-FDA approved CAR-T or BiTE product
2. Receiving Epcoritamab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-10-13 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
TempTraq's ability to measure axillary temperature in the intended use population. | Day 14
  Body temperature (degrees Celsius) data will be measured as a continuous variable via the TempTraq device and via standard-of-care oral thermometers.

SECONDARY OUTCOMES:
Lead time by which fevers can be detected using TempTraq compared to SOC interval oral thermometer measurements. | Day 14
  The times to first detection of fever, if applicable, will be measured for each patient using temperature data derived from the TempTraq device and standard-of-care oral thermometers. The mean time to first fever (i.e., temperature > 38 degrees Celsius), will be calculated and described for both the TempTraq device and standard-of-care oral thermometers.
VitalTraq's ability to measure blood pressure in the intended use population. | Day 14
  Determined by use of an equivalence test to test the hypothesis that there is no difference in the systolic and diastolic measurements using VitalTraq compared to SOC interval vitals measurements. The smallest tolerable differences in systolic and diastolic blood pressure are set to be 20 mmHg and 10 mmHg, respectively.
VitalTraq's ability to measure heart rate in the intended use population. | Day 14
  Determined by use of an equivalence test to test the hypothesis that there is no difference in the heart rate measurements using VitalTraq compared to SOC interval oral thermometer measurements. The smallest tolerable difference is set to be 10 beats per minute.
Patient's perspective on the burden of using TempTraq and VitalTraq. | Day 28
  The mean scores on individual questions in a post-intervention survey featuring 7-point Likert scale responses, where 1=strongly agree and 7=strongly disagree, will be calculated and described. A lower score indicates lower burden.
Lead time by which TempTraq and VitalTraq can detect grade 2 or higher Cytokine Release Syndrome (CRS) as compared to the standard of care. | Day 14
  The times to first detection of grade 2 or higher CRS, if applicable, will be measured for each patient using vitals data derived from the TempTraq and VitalTraq devices, as well as via standard-of-care vitals measurements. The mean time to first detection of grade 2 or higher CRS will be calculated and described for both the investigational devices and standard-of-care monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Chenyu Lin, MD, Principal Investigator — Duke University
Locations (1):
- Duke Blood Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No